CLINICAL TRIAL: NCT02152280
Title: A Clinical Trial of Danhong Injection in Treating Acute Ischemic Stroke
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Bozhiyin T&S Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V2.0
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — danhong; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Danhong Injection (Experimental): Danhong Injection 40 ml add 250 ml of 0.9% sodium chloride solution, injection intravenous drip, 1 time a day, for 10 days;
  Interventions: Drug: Danhong Injection
- Normal Saline (Placebo Comparator): 0.9% sodium chloride solution 40 ml add 250 ml of 0.9% sodium chloride solution, injection intravenous drip, 1 time a day, for 10 days.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Danhong Injection — Danhong Injection 40 ml add 250 ml of 0.9% sodium chloride solution, injection intravenous drip, 1 time a day, for 10 days.
  Arms: Danhong Injection
Drug: Normal Saline — 0.9% sodium chloride solution 40 ml add 250 ml of 0.9% sodium chloride solution, injection intravenous drip, 1 time a day, for 10 days;
  Arms: Normal Saline

SUMMARY:
Research topic.

* A clinical trial of Danhong injection in treating acute ischemic stroke .

Research purpose.

- To evaluate the efficacy and safety of Danhong injection in treating acute ischemic stroke by a randomized, double-blind, multi-center, placebo-controlled clinical trial.

Research design.

- A randomized, double-blind, multi-center, placebo-controlled clinical trial.

Subject crowd.

- Accord with standard of western medicine diagnosis of acute cerebral infarction, stroke and blood stasis type of traditional Chinese medicine syndrome differentiation.

Sample size. - Total sample size of 320 patients, experimental group, control group is equal to 1 to 1.

Interim analysis.

- Interim analysis will be performed when the total number of included patients up to half of the sample size ,160 cases, and according to the interim analysis results to estimate the sample size and adjust the project adaptively.

Course of treatment.

- 10 days.

Research endpoint.

- The 90th day after the medication for the first time.

Observation index.

1. General condition; the physical and chemical inspection related;
2. Efficacy check : mRS, BI, NIHSS;
3. Safety check: blood routine, urine routine, stool OB, liver function(ALT、AST), renal function (BUN, Cr), coagulation four indices（PT、APTT、TT、FIB), electrocardiogram.

Efficacy evaluation. 1. The main efficacy index: a. Percentage comparisons of two group patients of modified Rankin 0-2 grades on the 90th day.

Statistical analysis technique.

- Statistical analysis using SAS 9.2 system, all the statistical test adopted bilateral inspection, P value less than or equal to 0.05 will be considered a statistically significant difference.

DETAILED DESCRIPTION:
Research topic. - A clinical trial of Danhong injection in treating acute ischemic stroke .

Research purpose.

* To evaluate the efficacy and safety of Danhong injection in treating acute ischemic stroke by a randomized, double-blind, multi-center, placebo-controlled clinical trial.

Research design. - A randomized, double-blind, multi-center, placebo-controlled clinical trial.

Subject crowd. - Accord with standard of western medicine diagnosis of acute cerebral infarction, stroke and blood stasis type of traditional Chinese medicine syndrome differentiation.

Sample size.

- Total sample size of 320 patients, experimental group, control group is equal to 1 to 1.

Interim analysis.

- Interim analysis will be performed when the total number of included patients up to half of the sample size ,160 cases, and according to the interim analysis results to estimate the sample size and adjust the project adaptively.

Inclusion criteria.

1. Accord with the diagnostic criteria of cerebral infarction of "Guide of diagnosis and treatment of acute ischemic stroke in China" in 2010, and in the acute stage;
2. Accord with the stroke and blood stasis type;
3. Onset of acute ischemic stroke within 72 hours;
4. NIHSS grade ≥ 4;
5. Age ≥ 18;
6. signed the inform consent form.

Exclusion criteria.

1. Diagnosed with bleeding or other pathological brain disorders according to CT or MRI at baseline , such as vascular malformation, tumor, abscess or other common non ischemic cerebral disease (for multiple sclerosis);
2. Patients with hrombolysis or endovascular treatment;
3. Allergic constitution; the test drug allergy or its ingredients or elements allergy;
4. With severe liver function damage(ALT and AST level more than 1.5 times higher than normal);
5. With severe renal impairment (more than 1.5 times higher than normal amount of serum creatinine);
6. With severe cardiac insufficiency (cardiac function rating level III above);
7. Disabled patients of law (blind, deaf, dumb, mental retardation, mental disorder and physical disabilities caused by other reasons which affects the nerve function defect evaluation);
8. With bleeding tendency or had serious bleeding within 3 months;
9. Doubted or had alcohol and drug abuse history; Or who will lower the possibilities of enrollment or complicate the enrollment according to the investigaters' judgement;
10. Menstrual period women, pregnant women and lactating women, pregnancy test positive or recent family planning;
11. Who being in other clinical trials or had finished other clinical trials within 3 months.

    Dosage regimen.

    1. Experimental group: Danhong injection 40 ml add 250 ml of 0.9% sodium chloride solution, injection intravenous drip, 1 time a day, for 10 days; 2. Control group : 0.9% sodium chloride solution 40 ml add 250 ml of 0.9% sodium chloride solution, injection intravenous drip, 1 time a day, for 10 days.

    Course of treatment.
    * 10 days.

    Research endpoint.

    - The 90th day after the medication for the first time.

    Observation index.

<!-- -->

1. General condition; the physical and chemical inspection related;
2. Efficacy check : mRS, BI, NIHSS;
3. Safety check: blood routine, urine routine, stool OB, liver function(ALT、AST), renal function (BUN, Cr), coagulation four indices（PT、APTT、TT、FIB), electrocardiogram.

Observation point.

1. The physical and chemical inspection related and electrocardiogram observed at the enrollment time;
2. General condition and efficacy index observed on the 10th ,90th after the medication for the first time;
3. Safety index observed on the 10th after the medication for the first time.

Efficacy evaluation.

1. The main efficacy index:

   1. Percentage comparisons of two group patients of modified Rankin 0-2 grades on the 90th day.
2. The secondary efficacy index:

   1. Mortality comparisons of two group patients on the 90th day;
   2. Percentage comparisons of two group patients of BI≥75 on the 90th day;
   3. NIHSS difference comparisons of two group on the 90th day;
   4. The proportion of new vascular events within 3 months (Ischemic stroke/hemorrhagic stroke/TIA/MI/vascular death).

Safety evaluation.

1. All-Cause mortality within 90 days :the death toll of all cause within 90 days/ the total number of each group × 100%;
2. Incidence of serious bleeding events (GUSTO definition, appendix 4), including fatal bleeding and symptomatic intracranial bleeding;
3. Incidence of moderate bleeding events (GUSTO definition, appendix 4);
4. Adverse events and serious adverse events reported by investigaters.

Statistical analysis technique.

- Statistical analysis using SAS 9.2 system, all the statistical test adopted bilateral inspection, P value less than or equal to 0.05 will be considered a statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

* Accord with the diagnostic criteria of cerebral infarction of "Guide of diagnosis and treatment of acute ischemic stroke in China" in 2010, and in the acute stage;
* Accord with the stroke and blood stasis type;
* Onset of acute ischemic stroke within 72 hours;
* NIHSS grade ≥ 4;
* Age ≥ 18;
* signed the inform consent form.

Exclusion Criteria:

* Diagnosed with bleeding or other pathological brain disorders according to CT or MRI at baseline , such as vascular malformation, tumor, abscess or other common non ischemic cerebral disease (for multiple sclerosis);
* Patients with hrombolysis or endovascular treatment;
* Allergic constitution; the test drug allergy or its ingredients or elements allergy;
* With severe liver function damage(ALT and AST level more than 1.5 times higher than normal);
* With severe renal impairment (more than 1.5 times higher than normal amount of serum creatinine);
* With severe cardiac insufficiency (cardiac function rating level III above)
* Disabled patients of law (blind, deaf, dumb, mental retardation, mental disorder and physical disabilities caused by other reasons which affects the nerve function defect evaluation);
* With bleeding tendency or had serious bleeding within 3 months;
* Doubted or had alcohol and drug abuse history; Or who will lower the possibilities of enrollment or complicate the enrollment according to the investigaters' judgement;
* Menstrual period women, pregnant women and lactating women, pregnancy test positive or recent family planning;
* Who being in other clinical trials or had finished other clinical trials within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Percentage comparisons of two groups of patients on the modified Rankin Scale 0-2 grades on the 90th day. | 0-90 day
  Percentage comparisons of two groups of patients on the modified Rankin Scale 0-2 grades on the 90th day.

CONTACTS AND LOCATIONS:
Overall Officials: Fang D Cai, doctor, Principal Investigator — Traditional Chinese medicine department of Zhongshan Hospital